CLINICAL TRIAL: NCT01489592
Title: Effect of Curcumin on Iron Metabolism in Healthy Volunteer
Acronym: CURHEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C11-14; 2011-001925-26 (EudraCT Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2013-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — turmeric extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- curcumin (Experimental): oral administration of 6g of curcumin
  Interventions: Drug: curcuma longa
- placebo (Placebo Comparator): oral administration of 12 sugar pill
  Interventions: Drug: curcuma longa

INTERVENTIONS:
Drug: curcuma longa — oral administration of 6 grams of curcumin

SUMMARY:
The purpose of this study is to determine the impact of curcumin, administrated orally, on iron metabolism in healthy volunteers. Iron metabolism will be describe by hepcidin expression that the investigators observed in vitro and serum hepcidin levels.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 et 25 Kg/m²
* Non smoker
* No swallowing disorders
* Normal clinical exam
* Normal ECG
* Normal values for routine biological tests : serum iron, transferrin saturation,, hemogram ferritin, C Reactive Protein, AST, ALT, HDL and LDL cholesterol, triglycerides
* No C282Y mutation within the HFE gene
* Affiliation to social security
* Written informed consent obtained

Exclusion Criteria:

* Chronic or evolutive disease
* Infection during the 7 days before each sequence
* Drug or alcohol (>30g) abuse
* Current treatment
* Known food allergy
* stay at altitude (> 1500m) in 2 months
* Positive serology for hepatitis B or C virus or HIV.
* Transfusion or blood donation during the last three months.
* Exclusion period on the healthy volunteer National File.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximal variation of serum hepcidin level after oral administration of curcumin | within 48 hours after administration of curcumin

SECONDARY OUTCOMES:
Plasmatic iron bioavailability | 30min, 1H, 2H, 3H, 4H, 6H, 8H, 12H, 24H et 48H
  Iron, ferritin, transferrin, transferrin saturation
Evaluation of the inhibitory activity of volunteers's serum on hepcidin expression by hepatocytes | 30min, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h
  In vitro:
  * the coculture model that we previously developed to analyze endogenous hepcidin expression, and
  * human hepatic cells line (HepG2) stimulated or not by IL-6 which governs the STAT3 pathway, transfected with gene reporter constructs containing hepcidin promoter.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique (CIC) , 2 rue Henri Le Guilloux , CHU Pontchaillou, Rennes, France

REFERENCES:
- [Background] Laine F, Laviolle B, Bardou-Jacquet E, Fatih N, Jezequel C, Collet N, Ropert M, Morcet J, Hamon C, Reymann JM, Loreal O. Curcuma decreases serum hepcidin levels in healthy volunteers: a placebo-controlled, randomized, double-blind, cross-over study. Fundam Clin Pharmacol. 2017 Oct;31(5):567-573. doi: 10.1111/fcp.12288. Epub 2017 May 7. PMID 28370178
- [Background] Fatih N, Camberlein E, Island ML, Corlu A, Abgueguen E, Detivaud L, Leroyer P, Brissot P, Loreal O. Natural and synthetic STAT3 inhibitors reduce hepcidin expression in differentiated mouse hepatocytes expressing the active phosphorylated STAT3 form. J Mol Med (Berl). 2010 May;88(5):477-86. doi: 10.1007/s00109-009-0588-3. Epub 2010 Feb 19. PMID 20169331
- [Background] Loreal O, Haziza-Pigeon C, Troadec MB, Detivaud L, Turlin B, Courselaud B, Ilyin G, Brissot P. Hepcidin in iron metabolism. Curr Protein Pept Sci. 2005 Jun;6(3):279-91. doi: 10.2174/1389203054065392. PMID 15974953
- [Background] Verga Falzacappa MV, Vujic Spasic M, Kessler R, Stolte J, Hentze MW, Muckenthaler MU. STAT3 mediates hepatic hepcidin expression and its inflammatory stimulation. Blood. 2007 Jan 1;109(1):353-8. doi: 10.1182/blood-2006-07-033969. Epub 2006 Aug 31. PMID 16946298
- [Background] Sharma RA, Euden SA, Platton SL, Cooke DN, Shafayat A, Hewitt HR, Marczylo TH, Morgan B, Hemingway D, Plummer SM, Pirmohamed M, Gescher AJ, Steward WP. Phase I clinical trial of oral curcumin: biomarkers of systemic activity and compliance. Clin Cancer Res. 2004 Oct 15;10(20):6847-54. doi: 10.1158/1078-0432.CCR-04-0744. PMID 15501961
- [Background] Vareed SK, Kakarala M, Ruffin MT, Crowell JA, Normolle DP, Djuric Z, Brenner DE. Pharmacokinetics of curcumin conjugate metabolites in healthy human subjects. Cancer Epidemiol Biomarkers Prev. 2008 Jun;17(6):1411-7. doi: 10.1158/1055-9965.EPI-07-2693. PMID 18559556